CLINICAL TRIAL: NCT02639338
Title: A Phase 3, Global, Multicenter, Randomized, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir/Velpatasvir/GS-9857 Fixed-Dose Combination for 8 Weeks and Sofosbuvir/Velpatasvir for 12 Weeks in Subjects With Chronic Genotype 3 HCV Infection and Cirrhosis
Brief Title: Safety and Efficacy of SOF/VEL/VOX FDC for 8 Weeks and SOF/VEL for 12 Weeks in Adults Chronic Genotype 3 HCV Infection and Cirrhosis
Acronym: POLARIS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-367-1173; 2015-002996-12 (EudraCT Number)
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C Virus Infection
Keywords: Chronic
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — sofosbuvir velpatasvir voxilaprevir drug combination; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SOF/VEL/VOX (Experimental): SOF/VEL/VOX tablet for 8 weeks
  Interventions: Drug: SOF/VEL/VOX
- SOF/VEL (Experimental): SOF/VEL tablet for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL/VOX — 400/100/100 mg FDC tablet administered orally once daily with food
  Other Names: GS-7977/GS-5816/GS-9857; Vosevi®
  Arms: SOF/VEL/VOX
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily without regard to food
  Other Names: GS-7977/GS-5816; Epclusa®
  Arms: SOF/VEL

SUMMARY:
The primary objective of this study is to evaluate the efficacy, safety, and tolerability of treatment with sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) fixed-dose combination (FDC) for 8 weeks and of treatment with sofosbuvir/velpatasvir (SOF/VEL) FDC for 12 weeks in participants naive to direct-acting antivirals (DAA) with chronic genotype 3 hepatitis C virus (HCV) infection and cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL at screening
* Chronic genotype 3 HCV infection (≥ 6 months)
* Presence of cirrhosis
* HCV treatment naive or treatment experienced with an interferon (IFN)-based regimen
* Use of protocol specified methods of contraception

Key Exclusion Criteria:

* Current or prior history of clinically significant illness that may interfere with participation in the study
* Screening ECG with clinically significant abnormalities
* Laboratory parameters outside the acceptable range at screening
* Pregnant or nursing female
* Chronic liver disease not caused by HCV
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2017-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (70):
- United States (30):
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Rialto, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Miami, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Bastrop, Louisiana
  - Baltimore, Maryland
  - Catonsville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Hillsborough, New Jersey
  - New York, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Fayetteville, North Carolina
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Nashville, Tennessee
  - San Antonio, Texas
  - Murray, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Australia (6):
  - Camperdown, New South Wales
  - Darlinghurst, New South Wales
  - Herston, Queensland
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Melbourne, Victoria
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brampton, Ontario
  - Toronto, Ontario
- France (15):
  - Bobigny
  - Clermont-Ferrand
  - Clichy
  - Créteil
  - Limoges
  - Lyon
  - Marseille
  - Montpellier
  - Nice
  - Orléans
  - Paris
  - Pessac
  - Rennes
  - Strasbourg
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Berlin
  - Bonn
  - Cologne
  - Frankfurt am Main
  - Hamburg
  - Hanover
- New Zealand (2):
  - Grafton, Auckland
  - Christchurch
- San Juan, Puerto Rico
- United Kingdom (5):
  - London
  - Manchester
  - Nottingham
  - Oxford
  - Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/about/ethics-and-code-of-conduct/policies.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/about/ethics-and-code-of-conduct/policies

REFERENCES:
- [Result] Foster GR, Thompson AJ, Ruane PJ, Borgia SM, Dore G, Workowski K, et al. A Randomized Phase 3 Trial of Sofosbuvir/Velpatasvir/Voxilaprevir for 8 Weeks and Sofosbuvir/Velpatasvir for 12 Weeks for Patients with Genotype 3 HCV Infection and Cirrhosis: The POLARIS-3 Study [Abstract 258]. J Hepatology 2016;63 (1S):135A
- [Result] Jacobson IM, Lawitz E, Gane EJ, Willems BE, Ruane PJ, Nahass RG, Borgia SM, Shafran SD, Workowski KA, Pearlman B, Hyland RH, Stamm LM, Svarovskaia E, Dvory-Sobol H, Zhu Y, Subramanian GM, Brainard DM, McHutchison JG, Brau N, Berg T, Agarwal K, Bhandari BR, Davis M, Feld JJ, Dore GJ, Stedman CAM, Thompson AJ, Asselah T, Roberts SK, Foster GR. Efficacy of 8 Weeks of Sofosbuvir, Velpatasvir, and Voxilaprevir in Patients With Chronic HCV Infection: 2 Phase 3 Randomized Trials. Gastroenterology. 2017 Jul;153(1):113-122. doi: 10.1053/j.gastro.2017.03.047. Epub 2017 Apr 5. PMID 28390869

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Asia Pacific. The first participant was screened on 23 December 2015. The last study visit occurred on 02 January 2017.
Pre-assignment Details: 315 participants were screened.
Groups:
- SOF/VEL/VOX 8 Weeks: Sofosbuvir/Velpatasvir/Voxilaprevir (Vosevi®; SOF/VEL/VOX) (400/100/100 mg) fixed dose combination (FDC) tablet orally once daily with food for 8 weeks
- SOF/VEL 12 Weeks: Sofosbuvir/Velpatasvir (Epclusa®; SOF/VEL) (400/100 mg) FDC tablet orally once daily without regard to food for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Started | 110 | 110
Completed | 106 | 105
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrew Consent | 1 | 2
Not completed — Death | 1 | 0
Not completed — Randomized but Not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug
Groups:
- SOF/VEL/VOX 8 Weeks: SOF/VEL/VOX (400/100/100 mg) tablet orally once daily with food for 8 weeks
- SOF/VEL 12 Weeks: SOF/VEL (400/100 mg) tablet orally once daily without regard to food for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks | Total
Number analyzed (Participants) | 110 | 109 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8.5) | 55 (8.4) | 55 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 26 | 62
  Male | 74 | 83 | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 100 | 97 | 197
  Asian | 8 | 9 | 17
  American Indian or Alaska Native | 1 | 1 | 2
  Black or African American | 0 | 1 | 1
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 101 | 101 | 202
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 3 | 2 | 5
  Canada | 16 | 18 | 34
  United States | 50 | 46 | 96
  United Kingdom | 7 | 8 | 15
  Australia | 10 | 16 | 26
  France | 15 | 10 | 25
  Germany | 9 | 9 | 18
IL28b Status [Count of Participants; unit: Participants]
  CC | 41 | 52 | 93
  CT | 57 | 44 | 101
  TT | 12 | 13 | 25
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.0 (0.80) | 6.3 (0.63) | 6.2 (0.73)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 40 | 28 | 68
  ≥ 800,000 IU/mL | 70 | 81 | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all randomized/enrolled participants who took at least 1 dose of the study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL/VOX 8 Weeks: SOF/VEL/VOX (400/100/100 mg) FDC tablet orally once daily with food for 8 weeks
- SOF/VEL 12 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily without regard to food for 12 weeks
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 110 | 109
percentage of participants | 96.4 [91.0 to 99.0] | 96.3 [90.9 to 99.0]
Statistical Analysis 1: Comparison: SOF/VEL/VOX 8 Weeks; Test type: Superiority — The p-value is obtained from the 2-sided exact 1-sample binomial test for the superiority over the performance goal of 83%; p < 0.001, Binomial Test — The reported p-value was calculated. The statistical test was performed in SOF/VEL for 12 weeks at 0.05 significance level if and only if the statistical test performed in SOF/VEL/VOX for 8 weeks was significant at 0.05 significance level
Statistical Analysis 2: Comparison: SOF/VEL 12 Weeks; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, 2-sided exact 1-sample binomial test — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinue Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 110 | 109
percentage of participants | 0 | 0.9

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 110 | 109
percentage of participants
  SVR4 | 97.3 [92.2 to 99.4] | 97.2 [92.2 to 99.4]
  SVR24 | 96.4 [91.0 to 99.0] | 96.3 [90.9 to 99.0]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On Treatment
Time Frame: Weeks 1, 2, 4, 8 and 12
Population: Percentage of participants in Full Analysis Set with on-treatment data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 110 | 109
percentage of participants
  Week 1 | 17.3 [10.7 to 25.7] | 10.1 [5.1 to 17.3]
  Week 2: number analyzed (Participants) | 110 | 108
  Week 2 | 56.4 [46.6 to 65.8] | 50.9 [41.1 to 60.7]
  Week 4: number analyzed (Participants) | 110 | 108
  Week 4 | 87.3 [79.6 to 92.9] | 85.2 [77.1 to 91.3]
  Week 8: number analyzed (Participants) | 110 | 108
  Week 8 | 97.3 [92.2 to 99.4] | 99.1 [94.9 to 100.0]
  Week 12: number analyzed (Participants) | 0 | 107
  Week 12 |  | 100.0 [96.6 to 100.0]

5. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Weeks 1, 2, 4, 8 and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 110 | 109
log10 IU/mL
  Week 1: number analyzed (Participants) | 106 | 105
  Week 1 | -4.06 (0.716) | -4.09 (0.653)
  Week 2: number analyzed (Participants) | 109 | 107
  Week 2 | -4.60 (0.825) | -4.73 (0.783)
  Week 4: number analyzed (Participants) | 109 | 108
  Week 4 | -4.84 (0.789) | -5.00 (0.781)
  Week 8: number analyzed (Participants) | 107 | 108
  Week 8 | -4.90 (0.801) | -5.09 (0.832)
  Week 12: number analyzed (Participants) | 0 | 107
  Week 12 |  | -5.14 (0.630)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment), or
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 110 | 109
percentage of participants | 1.8 | 1.8

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Serious Adverse Events (participants affected / at risk) | 2/110 | 3/109
Other Adverse Events (participants affected / at risk) | 68/110 | 61/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX 8 Weeks (N=110) | SOF/VEL 12 Weeks (N=109)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX 8 Weeks (N=110) | SOF/VEL 12 Weeks (N=109)
Abdominal pain (Gastrointestinal disorders) | 9 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 17 | 5
Nausea (Gastrointestinal disorders) | 23 | 10
Vomiting (Gastrointestinal disorders) | 7 | 1
Fatigue (General disorders) | 28 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Headache (Nervous system disorders) | 27 | 32
Insomnia (Psychiatric disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years